CLINICAL TRIAL: NCT05171634
Title: Impact of Artificial Intelligence in Dysplasia Detection During Colonoscopy in Patients With Long-data Ulcerative Colitis: a Crossover Study
Brief Title: Artificial Intelligence and Dysplasia Detection in Ulcerative Colitis (CUDISIA Study)
Acronym: CUDISIA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana (Other)
Collaborators: University of Valencia (Other)
Responsible Party: Principal Investigator, Antonio López-Serrano, Chief of Endoscopy, Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana
Allocation: Non-Randomized | Model: Crossover | Masking: Double | Purpose: Screening
Other Study IDs: CEIm: 62.21
Record Dates: First submitted 2021-06-16; First posted 2021-12-29 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Ulcerative Colitis; Dysplasia
Keywords: Virtual chromoendoscopy; Artificial intelligence; iSCAN; Dysplasia
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Colonoscopy assisted by DiscoveryTM (Experimental)
  Interventions: Device: DiscoveryTM
- Virtual Colonoscopy with iSCAN (Active Comparator)
  Interventions: Device: iSCAN

INTERVENTIONS:
Device: DiscoveryTM — Colonoscopy assisted by an artificial intelligence system (DiscoveryTM).
  Arms: Colonoscopy assisted by DiscoveryTM
Device: iSCAN — Virtual colonoscopy assisted by iSCAN
  Arms: Virtual Colonoscopy with iSCAN

SUMMARY:
Prospective clinical study that analyzes the efficacy of colonoscopy assisted by an artificial intelligence system (DiscoveryTM) compared to virtual chromoendoscopy with iSCAN in the detection of colon dysplasia in patients with long-standing Ulcerative Colitis.

ELIGIBILITY:
Inclusion Criteria:

* Ulcerative Colitis confirmed by endoscopy and histology.
* Involvement 30% of the colonic surface (or any extent if concomitant with PSC).
* Duration of the disease >7 years (or any duration if concomitant with PSC).

Exclusion Criteria:

* Personal history of colorectal cancer or high-grade dysplasia.
* Previous colectomy (partial or complete).
* Coagulopathy that prevents biopsies or polypectomy.
* Colonoscopy performed in the previous 6 months.
* Pregnant or nursing women.
* Inadequate bowel preparation.
* Presence of endoscopic Ulcerative Colitis activity.
* Colonic stenosis and incomplete colonoscopy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-05-05 (Actual); Primary Completion 2021-05-18 (Actual); Study Completion 2021-05-18 (Actual)

PRIMARY OUTCOMES:
"Per lesion" dysplasia detection rate (DDR) | Immediately after the procedure.
  Proportion of dysplastic lesions in relation to all the lesions analyzed that were detected by Artificial Intelligence System (DiscoveryTM) or Virtual chromoendoscopy with iSCAN in patients with long-standing Ulcerative Colitis who undergo surveillance colonoscopy.
"Per patient" dysplasia detection rate (DDR) | Immediately after the procedure.
  Proportion of patients with dysplastic lesions in relation to all the patients with long-standing Ulcerative Colitis included in the study detected by Artificial Intelligence System (DiscoveryTM) or Virtual chromoendoscopy with iSCAN.

CONTACTS AND LOCATIONS:
Locations (1):
- Antonio López-Serrano, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lopez-Serrano A, Voces A, Lorente JR, Santonja FJ, Algarra A, Latorre P, Del Pozo P, Paredes JM. Artificial intelligence for dysplasia detection during surveillance colonoscopy in patients with ulcerative colitis: A cross-sectional, non-inferiority, diagnostic test comparison study. Gastroenterol Hepatol. 2025 Feb;48(2):502210. doi: 10.1016/j.gastrohep.2024.502210. Epub 2024 May 11. English, Spanish. PMID 38740327
- See also: Related Info — https://www.elsevier.es/es-revista-gastroenterologia-hepatologia-14-linkresolver-artificial-intelligence-for-dysplasia-detection-S0210570524001687